CLINICAL TRIAL: NCT05149378
Title: Venetoclax Based Regimen for the Treatment of Relapsed or Refractory T-cell Acute Lymphoblastic Leukemia
Brief Title: Venetoclax Based Regimen for R/R T-ALL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Jining Medical University (Other); The Second People's Hospital of Huai'an (Other); The First Affiliated Hospital of Bengbu Medical University (Other); Affiliated Hospital of Nantong University (Other); Suzhou Hospital of Traditional Chinese Medicine (Other); The First Affiliated Hospital of Anhui Medical University (Other); Southern Medical University, China (Other); Nanyang Central Hospital of Henan Province (Unknown); Canglang Hospital of Suzhou (Unknown)
Responsible Party: Principal Investigator, Sheng-Li Xue, MD, Prof., The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZRTALL01
Record Dates: First submitted 2021-11-25; First posted 2021-12-08 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Acute T-Lymphocytic Leukemia
Keywords: venetoclax; relapse; refractory
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venetclax combined with azacitidine (Experimental): Relapsed or refractroy acute lymphoblastic leukemia patients reveive venetclax combined with azacitidine regimen treatment.
  Interventions: Drug: Venetoclax combined with azacitidine regimen

INTERVENTIONS:
Drug: Venetoclax combined with azacitidine regimen — Venetoclax orally once daily (100 mg d1, 200 mg d2, 400 mg d3-21); azacitidine 75 mg/m2 subcutaneously once daily on days 1-7 .

SUMMARY:
This study is to investigate the therapeutic efficacy and side effect of venetoclax based regimen for relapsed or refractroy T cell acute lymphoblastic leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 15 and ≤ 70 years.
2. Patients diagnosed with T-ALL/LBL according to 2017 WHO lymphoid malignant disease diagnosis standard.
3. Patients with T-ALL/LBL must meet one of the following criteria, A or B.

   A: Refractory T-ALL/LBL disease was defined as follows: Failure to achieve CR at the end of induction.

   B: Relapsed T-ALL/LBL disease was defined as follows: Reappearance of blasts in the blood or bone marrow (>5%) or in any extramedullary site after a CR.
4. ECOG performance status score less than 3.
5. Expected survival time >3 months.
6. Patients without serious heart, lung, liver, or kidney disease.
7. Ability to understand and voluntarily provide informed consent.

Exclusion Criteria:

1. Patients who are allergic to the study drug or drugs with similar chemical structures.
2. Pregnant or lactating women, and women of childbearing age who do not want to practice effective methods of contraception.
3. Active infection.
4. Active bleeding.
5. Patients with new thrombosis, embolism, cerebral hemorrhage, or other diseases or a medical history within one year before enrollment.
6. Patients with mental disorders or other conditions whereby informed consent cannot be obtained and where the requirements of the study treatment and procedures cannot be met.
7. Liver function abnormalities (total bilirubin > 1.5 times the upper limit of the normal range, ALT/AST > 2.5 times the upper limit of the normal range or patients with liver involvement whose ALT/AST > 1.5 times the upper limit of the normal range), or renal anomalies (serum creatinine > 1.5 times the upper limit of the normal value).
8. Patients with a history of clinically significant QTc interval prolongation (male > 450 ms; female > 470 ms), ventricular heart tachycardia and atrial fibrillation, II-degree heart block, myocardial infarction attack within one year before enrollment, and congestive heart failure, and patients with coronary heart disease who have clinical symptoms and requiring drug treatment.
9. Surgery on the main organs within the past six weeks.
10. Drug abuse or long-term alcohol abuse that would affect the evaluation results.
11. Patients who have received organ transplants (excepting bone marrow transplantation).
12. Patients not suitable for the study according to the investigator's assessment.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | At the end of Cycle 1 (each cycle is 21 days)
  The overall response (complete remission, complete remission with incomplete blood count recovery) rate achieved after one or two courses (21 days) induction therapy by venetoclax combined azacitidine regimen.
Complete Remission Rate (CRR) | At the end of Cycle 1 (each cycle is 21 days)
  The complete remission rate achieved after one or two courses (21 days) induction therapy by venetoclax combined azacitidine regimen.

SECONDARY OUTCOMES:
Overall survial (OS) | 1 year
  It is measured from the date of entry into this trial to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.
Relapse-Free Survival (RFS) | 1 year
  It is measured from the date of entry into this trial to the date of hematologic relapse or death from any cause.
Adverse events in hematological system | 1 month
  Record of adverse events in hematological system during and after designed venetoclax combined azacitidine regimen induction.
Adverse events in other organs or systems | 1 month
  Record of adverse events in other organs or systmes during and after designed venetoclax combined azacitidine regimen induction.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cao HY, Zhang H, Zhang Y, Hu XH, Yang L, Yang YL, Zhang YM, Wu B, Huang ZQ, Huang R, Wang RJ, Wan CL, Wu DP, Dai HP, Xue SL. Venetoclax plus azacitidine in relapsed or refractory T-cell acute lymphoblastic leukaemia: a multicentre, single-arm, phase 2 trial. Lancet Haematol. 2025 Dec;12(12):e946-e955. doi: 10.1016/S2352-3026(25)00284-4. PMID 41338863